CLINICAL TRIAL: NCT06823453
Title: Reducing Overdose and Substance Use-related Stigma on Chicago's West Side by Training Non-substance-using Friends and Family Members of People Who Use Opioids to Be Harm Reduction Champions
Brief Title: Reducing Overdose and Substance Use-related Stigma by Training Non-substance-using Friends and Family Members of People Who Use Opioids to Be Harm Reduction Champions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CE003666 (NIH); R01CE003666 (NIH)
Record Dates: First submitted 2025-02-03; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Opioid Overdose Prevention; People Who Use Opioids/People With Opioid Use Disorder (OUD); Reduction of Substance Use-related Stigma; Non-substance-using People With a Friend or Family Member Who Uses Opioids; Peer Harm Reduction Support Champions
Keywords: opioid overdose prevention; drug overdose prevention; overdose prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Harm Reduction Support Champion Intervention (Active Comparator): This intervention will recruit non-substance-using friends and family members of people who use opioids and live on the West side of Chicago, educate them on harm reduction (HR) tools and services, and train them to become peer HR support champions. They will be asked to recruit one friend or family member who uses opioids to the study, who will also be provided with an educational training on overdose risk reduction and available HR tools and services. The intervention will then facilitate a counselor-led initial conversation between peer HR support champions and their friend or family member who uses opioids, to help establish HR-related support, and will provide all participants with naloxone and fentanyl test strip kits. This intervention will not only provide another mechanism through which people who use opioids can access HR tools and services, thereby reducing logistical barriers to access and preventing overdose, but it should also reduce stigma and increase social support.
  Interventions: Behavioral: Peer Harm Reduction Support Champion Intervention
- Non-equivalent comparison group of PWUD with some recent access to harm reduction services (No Intervention): A non-equivalent comparison group will be recruited of people who use drugs (PWUD) who have recently (in the last six months) accessed harm reduction services from one of the study's community partners.

INTERVENTIONS:
Behavioral: Peer Harm Reduction Support Champion Intervention — This intervention will recruit non-substance-using friends and family members of people who use opioids and live on the West side of Chicago, educate them on harm reduction (HR) tools and services, and train them to become peer HR support champions. They will be asked to recruit one friend or family member who uses opioids to the study, who will also be provided with an educational training on overdose risk reduction and available HR tools and services. The intervention will then facilitate a counselor-led initial conversation between peer HR support champions and their friend or family member who uses opioids, to help establish HR-related support, and will provide all participants with naloxone and fentanyl test strip kits. This intervention will not only provide another mechanism through which people who use opioids can access HR tools and services, thereby reducing logistical barriers to access and preventing overdose, but it should also reduce stigma and increase social support.
  Arms: Peer Harm Reduction Support Champion Intervention

SUMMARY:
Fatal opioid overdoses are more frequent among populations with low access to harm reduction (HR) services and with high substance use-related stigma (which is a major barrier to accessing HR services). One such population is older adults who use drugs (PWUD) on the West side of Chicago. Over 34% of Chicago's opioid-related EMS responses in 2023 were located in communities on the West side, but older adults in these communities access HR services at low rates, likely due to stigma and other barriers. To help address these barriers and increase HR service access among this population, the proposed clinical trial will evaluate a novel intervention that will recruit non-substance-using friends and family members of people who use opioids and live on the West side of Chicago, educate them on HR tools and services, and train them to become peer HR support champions. They will be asked to recruit one friend or family member who uses opioids to the study, who will also be provided with an educational training on overdose risk reduction and available HR tools and services. The intervention will then facilitate a counselor-led initial conversation between peer HR support champions and their friend or family member who uses opioids to help establish HR support, and provide all participants with naloxone and fentanyl test strip kits. This intervention will not only provide another mechanism through which PWUD can access HR tools and services, thereby reducing logistical barriers, but should also reduce stigma and increase social support by facilitating and normalizing open conversations about HR between PWUD and their non-PWUD HR support champions. Participants of a previous focus group conducted by the Investigators among West side PWUD thought this intervention would be helpful, said they would be willing to participate in it, and said they knew someone who could participate as their non-PWUD peer HR support champion. To facilitate recruitment of older adults, the Investigative Team will work with local faith-based and service organizations and educate them about the importance of HR. The intervention's efficacy will be evaluated for a) increasing uptake/use of HR services, b) decreasing overdose frequency, and c) decreasing stigma and other barriers to accessing HR services, both i) by examining change over time among intervention participants, and ii) by using propensity-score matching methods to compare outcomes between intervention participants and a comparison group of PWUD who have recently accessed HR services from one of the study's community partners (Community Outreach Intervention Projects or West Side Heroin and Opioid Task Force).

DETAILED DESCRIPTION:
Study Overview. The goal of the proposed study is to conduct a clinical trial to a) evaluate the feasibility and acceptability of and b) evaluate the efficacy of a peer harm reduction support champion intervention that is designed to increase access to harm reduction tools and services and prevent opioid overdose by increasing social support, decreasing substance use-related stigma, and addressing barriers to accessing harm reduction tools and services. This novel intervention will recruit non-substance-using friends and family members (i.e., "peers") of people who use opioids and live on the West side of Chicago, educate them on harm reduction tools and services, and train them to become peer harm reduction support champions. They will be asked to recruit one friend or family member who uses opioids to the study, who will also be provided with an educational training on overdose risk reduction and available harm reduction tools and services. The intervention will then facilitate a counselor-led initial conversation between peer harm reduction support champions and their friend or family member who uses opioids, to help establish harm reduction-related support, and will provide all participants with naloxone and fentanyl test strip kits. This intervention will not only provide another mechanism through which people who use drugs (PWUD) can access harm reduction tools and services, thereby reducing logistical barriers to access and preventing overdose, but it should also reduce stigma and increase social support by facilitating and normalizing open conversations about harm reduction between PWUD and their non-PWUD harm reduction support champions.

Intervention participants will be recruited to the study using two strategies: 1) non-PWUD peers will be directly recruited to be trained as harm reduction support champions, and then asked to recruit their peer who uses drugs (i.e., PWUD partner) who they will provide with support; and 2) PWUD will be directly recruited - with an emphasis on trying to recruit PWUD who have not recently accessed harm reduction services (though this will not be an eligibility requirement) - to the intervention, and then asked to recruit a non-PWUD peer who is willing to offer them harm reduction-related support. Separate recruitment will be conducted of comparison group participants (specifically, a comparison group of PWUD who have recently accessed harm reduction services from one of the study's community partners). Participants will either be recruited to the intervention to participate with their peer partners, as described above, or they will be recruited to the non-equivalent comparison group of people who use opioids who have recently accessed harm reduction services from one of the study's community partners (i.e., there will be no random assignment). To facilitate recruitment of older adults to the intervention, the Investigative Team will work with local faith-based organizations and service-providing organizations in the Austin and Garfield Park communities. This effort will be led by two faith-based consultants (the Director of Community Relations from Breakthrough Urban Ministries; and a local pastor who is also Director of the West Side Heroin and Opioid Task Force) who will help the study team build relationships with faith-based organizations and service-providing organizations and educate them about the importance of HR. Study recruitment fliers will be disseminated through these organizations. All participants will be interviewed and assessed at baseline, and will also be asked to complete 1-month, 3-month, and 6-month follow-up interviews. The intervention's efficacy will be evavluated for a) increasing uptake/use of harm reduction services, b) decreasing overdose frequency, and c) decreasing stigma and other barriers to accessing HR services, both i) by examining change over time among intervention participants, and ii) by using propensity-score matching quasi-experimental methods to compare outcomes between intervention participants and comparison group participants.

Recruitment Coupons. All recruitment of participants' peer partners in the intervention condition will occur via the distribution of recruitment coupons by participants. Coupons will contain unique, confidential alpha-numeric codes which will not contain any identifying information about the participant, but which will be used to link participants' peer partners to them for analytic purposes. To protect participants' privacy, coupons will state only that the study is about "community health." Coupon design and language will be reviewed and approved by UIC's IRB.

Number and Characteristics of Participants to Be Enrolled. A planned total of 600 human subjects will be involved in the proposed research. Of these, 300 will be intervention participants, and 300 will be non-equivalent comparison group participants. Of the 300 intervention participants, 150 will be people who use opioids, and 150 will be non-substance-using friends and family members (i.e., "peers") of the 150 participants who use opioids, who will be trained to become peer harm reduction support champions. The 300 non-equivalent comparison group participants will be people who use drugs (PWUD) - specifically, opioids - who have recently accessed harm reduction services from one of the study's community partners: Community Outreach Intervention Projects (COIP) or West Side Heroin and Opioid Task Force (WSHOTF). The purpose of recruiting a comparison group of 300 PWUD to compare to the 150 intervention participants who are PWUD is to ensure adequate matching of intervention group and comparison group participants on socioeconomic and demographic characteristics for propensity-score matching analysis.

Baseline Quantitative Interviews. All participants will be interviewed about their sociodemographic and socioeconomic characteristics, knowledge of harm reduction tools and services, experiences of substance use-related stigma and social support, perception of the level of substance use-related stigma in their communities, and depression and anxiety in the last month. Intervention participants will be asked about their relationship (type, length, and closeness) to their peer partner that is enrolled in the intervention. All PWUD participants (in the intervention group and comparison group) will be asked about their drug use behaviors (including how often they use drugs alone) and overdose experiences during the last three months, their access to and use of harm reduction tools and services and/or drug treatment in the last three months, and any barriers they have experienced to accessing or using these services. Audio computer-assisted self-interviewing (ACASI) will be used to ask questions about sensitive topics such as drug use behaviors, such that participants will not have to answer these questions out loud.

Follow-Up Quantitative and Qualitative Interviews. Participants will be asked to return to complete follow-up interviews approximately 1 month, 3 months, and 6 months after they have completed intervention activities (for intervention participants), or after their baseline interviews (for comparison group participants). At each time point, follow-up interviews will ask all participants about their knowledge of harm reduction tools and services, experiences of substance use-related stigma and social support, perception of the level of substance use-related stigma in their communities, and depression and anxiety in the last month. Follow-up interviews for PWUD participants (in the intervention group and comparison group) will also ask about participants' drug use behaviors, overdose experiences, access to and use of harm reduction tools and services, and barriers to accessing or using such services during the period between the last interview and each follow-up interview. Follow-up interviews for intervention participants will also ask about how often participants discussed harm reduction with their peer partner, and what services they helped their partner access (for non-PWUD) or accessed with the help of their partner (for PWUD). This will include whether the non-PWUD partner was intentionally present or available while the PWUD partner was using drugs, in order to avoid the PWUD partner using drugs alone. Intervention participants will also be asked to rate the acceptability, appropriateness, and feasibility of the intervention during the 1-month and 6-month follow-up interviews, and will ask questions to monitor for any distress or relationship strain between peer pairs at every follow-up interview. Any negative experiences reported will be followed up and evaluated as potential Adverse Events (see DSMP).

Brief (30 minutes or less) qualitative interviews will be conducted with intervention participants at each follow-up time point, and immediately following the counselor-facilitated harm reduction support discussion between peer pairs (a component of the intervention), to obtain participant feedback on the intervention. These qualitative interviews will include the following topics: feasibility and acceptability of each component of the intervention (recruiting peers, educational training, counselor-facilitated conversations, and receipt of naloxone and fentanyl test strip kits); participants' reactions to being recruited by their peer, or the reactions of the peer(s) they tried to recruit; participant comfort with helping or being helped with access to specific different harm reduction tool, services, and overdose prevention strategies; perceptions of productiveness of counselor-facilitated conversation with peer; conversational ease or awkwardness during counselor-facilitated conversation; anticipated comfort with having future conversations about HR services with peers; and any distress or discomfort experienced during any intervention component.

Participant Locator Forms. All participants will be asked to complete a locator form at the time of their baseline interviews, in order to obtain information to use to contact participants for follow-up interviews. Participants will be informed during the consent process about this follow-up component, and consent forms will obtain permission to contact them again for their 1-month, 3-month, and 6-month follow-up interviews. Locator forms will include the participants' own contact information, as well as information about other individuals who might be able to help locate the participant if direct attempts are unsuccessful.

Outcomes to Be Compared between Study Arms to Evaluate Intervention Efficacy. Outcomes to be compared between intervention and comparison group arms to evaluate the efficacy of the peer harm reduction support champion intervention are: uptake/use of harm reduction tools and services, overdose frequency, substance use-related stigma, barriers to accessing harm reduction services, and perceptions of social support.

ELIGIBILITY:
Eligibility Criteria for Non-PWUD (i.e., people who do not use drugs) Peer Intervention Participants, to Be Trained as Harm Reduction Support Champions. 1) Non-PWUD peers recruited directly to the study (i.e., not by a PWUD peer partner) will be eligible to participate in the intervention arm of the study if they live in Chicago, know someone at least 18 years of age who lives on the West side of Chicago who currently uses opioids (to the best of their knowledge), state that they are interested in learning how to offer social support and practical support to that person, report that they have not used "hard" drugs (drugs other than alcohol or marijuana) recreationally in the last year, are at least 18 years of age, and state that they and the person they want to support are able to be interviewed in English and/or Spanish. 2) Non-PWUD peers recruited to the intervention arm of the study by a study participant they know who uses drugs will be eligible to participate in the intervention if they live in Chicago, report that they have not used "hard" drugs (drugs other than alcohol or marijuana) recreationally in the last year, state that they are willing to learn how to support their peer who uses drugs, are at least 18 years old, and are able to be interviewed in English and/or Spanish.

Eligibility Criteria for PWUD Intervention Participants (i.e., intervention participants who use drugs). 1) People who use drugs (PWUD) recruited directly to the intervention arm of the study (i.e., not by a non-PWUD peer partner) by West Side Heroin and Opioid Task Force or snowball sampling will be eligible to participate in the intervention if they live on the West side of Chicago, report that they currently use opioids (i.e., in the last week), know at least one person living in Chicago who has not used opioids in the last year and who they are willing to try to recruit to the study as someone who might be willing to offer them harm reduction support, are at least 18 years old, and are able to be interviewed in English and/or Spanish. 2) PWUD recruited to the intervention arm of the study by their non-PWUD peers who are enrolled in the study will be eligible to participate in the intervention group if they live in Chicago, have a study recruitment coupon from a non-PWUD participant, report that they currently use opioids (i.e., in the last week), state that they are willing to learn how their peer might be able to support them, are at least 18 years of age, and are able to be interviewed in English and/or Spanish.

Eligibility Criteria for Non-equivalent Comparison Group Participants. Comparison group participants will be eligible to participate in the comparison arm of the study if they report currently using opioids (i.e., in the last week), have accessed harm reduction services from one of the study's community partners (Community Outreach Intervention Projects; or West Side Heroin and Opioid Task Force) in the last six months, are at least 18 years old, and are able to speak English and/or Spanish. These individuals who are recruited to the comparison group will not be eligible to participate in the intervention unless they are given a recruitment coupon by a non-PWUD peer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Overdose Frequency and Experiences | baseline, 1 month, 3 months, 6 months
  Overdose frequency and experiences will be measured using participant self-report on items used by the Investigators in previous studies of PWUD. Items will ask about the number of overdoses participants experienced in the last three months (at baseline) and since the last interview (for follow-up). For each overdose reported, items will ask whether the participant was alone, whether naloxone was used, whether first responders were called, and whether an emergency room visit occurred. Participants will also be asked to report on whether they were present while someone else overdosed, and if so, whether they or someone else used naloxone.
Number of Types of Harm Reduction Services Accessed | baseline, 1 month, 3 months, 6 months
  This will be measured using participant self-report. Participants will be asked about their harm reduction service access and use in the last three months (at baseline) and since the last interview (for follow-up). Specifically, participants will be asked to report on how many times they accessed or received naloxone and fentanyl test strip kits, used fentanyl test strip kits, used "never use alone" hotlines, used "safe spaces" to use drugs or to experience withdrawal, used syringe service programs, tested for HIV or HCV, accessed medication for opioid use disorder, and accessed other types of drug treatment. A composite score will be computed reflecting the number of types of harm reduction tools and services accessed, which will be a count of all service/tool types accessed or used.
Frequency of Access to Harm Reduction Tools and Services | baseline, 1 month, 3 months, 6 months
  This will be measured using participant self-report. Participants will be asked about their harm reduction service access and use in the last three months (at baseline) and since the last interview (for follow-up). Specifically, participants will be asked to report on how many times they accessed or received naloxone and fentanyl test strip kits, used fentanyl test strip kits, used "never use alone" hotlines, used "safe spaces" to use drugs or to experience withdrawal, used syringe service programs, tested for HIV or HCV, accessed medication for opioid use disorder, and accessed other types of drug treatment. A composite score will be computed reflecting frequency of access to these tools and services, which will be a sum of the total number of times each participant used any of the harm reduction tools and services above.

SECONDARY OUTCOMES:
Barriers to Harm Reduction Services (Number of Types of Barriers) | baseline, 1 month, 3 months, 6 months
  Barriers to harm reduction services will be measured using participant self-report on items used by the Investigators in previous studies of PWUD. Participants will be asked how many times they have wanted to access harm reduction tools or services but were not able to do so, which tools or services they were unable to access, and what prevented them from accessing them. Specifically, participants will be asked about naloxone and fentanyl test strip unavailability, transportation barriers, time of day/scheduling challenges (i.e., services were not available or open at the specific time of day/day of week needed), and whether anticipated stigma/fear of stigma was a barrier to seeking/obtaining services or tools. The total number of types of barriers experienced for each participant will be computed.
Barriers to Harm Reduction Services (Frequency of Experiencing Barriers) | baseline, 1 month, 3 months, 6 months
  Barriers to harm reduction services will be measured using participant self-report on items used by the Investigators in previous studies of PWUD. Participants will be asked how many times they have wanted to access harm reduction tools or services but were not able to do so, which tools or services they were unable to access, and what prevented them from accessing them. Specifically, participants will be asked about naloxone and fentanyl test strip unavailability, transportation barriers, time of day/scheduling challenges (i.e., services were not available or open at the specific time of day/day of week needed), and whether anticipated stigma/fear of stigma was a barrier to seeking/obtaining services or tools. The sum of the number of times participants experienced any of the barriers above will be computed.
Substance Use-related Stigma (Individual Experiences of Stigma) | baseline, 1 month, 3 months, 6 months
  Participants' experiences of substance use-related stigma will be measured using the Substance Use Stigma Mechanisms Scale (SU-SMS).
Substance Use-related Stigma (Perception of Community-Level Stigma) | baseline, 1 month, 3 months, 6 months
  Perceptions of substance use-related stigma in participants' communities will be measured by adapting a 7-item measure developed by PI Williams and the SIZE research team such that it will ask how likely respondents think people who use drugs are to experience stigmatizing behavior from people in their community.
Peer Facilitation of Harm Reduction Service Access (Discussions about Harm Reduction) | baseline, 1 month, 3 months, 6 months
  Peer support and facilitation of harm reduction service access will be measured using participant self-report. All intervention participants will be asked at each follow-up interview how many times (since the last interview) they discussed harm reduction with their peer partner.
Peer Facilitation of Harm Reduction Service Access (Frequency of Collaborative or Peer-Facilitated Access) | baseline, 1 month, 3 months, 6 months
  Peer support and facilitation of harm reduction service access will be measured using participant self-report. PWUD who receive the intervention will be asked at each follow-up interview to report how many times (since the last interview) they accessed harm reduction services with the help of their partner (for PWUD). This will include how many times their non-PWUD partner was ever intentionally present or available while the PWUD partner was using drugs, in order to help them avoid using alone. Non-PWUD peers will be asked at each follow-up interview to report how many times they helped their partner access harm reduction services since the last interview. This will include how many times they were intentionally present or available while the PWUD partner was using drugs, in order to help the PWUD partner avoid using alone.
Social Support | baseline, 1 month, 3 months, 6 months
  General quality of social support will be collected for all participants, using the 24-item Social Provisions Scale (SPS), which assesses quality of social support received and/or provided to others, and has been used with good internal consistency among PWUD.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie D. Williams, Ph.D., Principal Investigator — University of Illinois Chicago
Locations (1):
- Community Outreach Intervention Projects (COIP), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
In keeping with the goal of maximizing data sharing, the Investigators will deposit de-identified project data in openICPSR©. The de-identified data will be preserved as-is and available to data users at no cost for a minimum of ten years. openICPSR© requires that data users must be granted approval for access.
  All data will be completely de-identified to ensure participant confidentiality. Users of the public use data will be required to register with ICPSR and agree to its Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, by prohibiting attempts to identify study participants, and by requiring immediate reporting of attempts to identify study participants, and by requiring immediate reporting of any disclosure of study participant identity. Data users will also be required to agree not to share or redistribute any data downloads.
Supporting Information: Study Protocol
Time Frame: Within 12 months of the publication of the set of papers that address the main specific aims of this study, all data will be compiled in a standard statistical software and available for open access. The data will be available for a minimum of ten years.
Access Criteria: OpenICPSR© is a secure repository for storing and sharing social and behavioral science research data. To ensure confidentiality and to protect sensitive data, openICPSR© reviews all data to assess disclosure risk and to determine the level of access (open or restricted). Additionally, openICPSR© requires that data users must be granted approval for access, and in cases of restricted data, allows access only via controlled virtual labs. Users of the public use data will be required to register with ICPSR and agree to its Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, by prohibiting attempts to identify study participants, and by requiring immediate reporting of any disclosure of study participant identity. Data users will also be required to agree not to share or redistribute any data downloads.
URL: https://www.openicpsr.org/openicpsr/